CLINICAL TRIAL: NCT03856372
Title: Postmastectomy Hypofractionated Versus Conventional Fractionated Radiotherapy in High Risk Breast Cancer: a Phase III Randomized Clinical Trial
Brief Title: Hypofractionated Vs Conventional Fractionated Postmastectomy Radiotherapy for High Risk Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jinli Ma, Associate Professor of department of radiation oncology, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FDRT-BC008
Record Dates: First submitted 2019-02-20; First posted 2019-02-27 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Breast Cancer
Keywords: Postmastectomy Hypofractionated Adjuvant Radiotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiation Dose Hypofractionation; Congresses as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypofractionated (Experimental): 42.5 Gy / 16 fractions, 2.66 Gy per fraction, 5 fractions weekly
  Interventions: Radiation: Hypofractionated
- Conventional (Active Comparator): 50 Gy / 25 fractions, 2.00 Gy per fraction, 5 fractions weekly
  Interventions: Radiation: Conventional

INTERVENTIONS:
Radiation: Hypofractionated — daily fractions, five fractions per week.
  Other Names: Experimental Arm
  Arms: Hypofractionated
Radiation: Conventional — daily fractions, five fractions per week.
  Other Names: Standard Arm
  Arms: Conventional

SUMMARY:
The study was designed to investigate whether hypofractionated adjuvant radiotherapy is noninferior to conventionally fractionated adjuvant radiotherapy in terms of efficacy and toxicities for high risk breast cancer patients treated with mastectomy

DETAILED DESCRIPTION:
The randomization is between 50 Gy / 25 fractions and 42.5 Gy/16 fractions, 5 fractions weekly.

Eligible breast cancer patients with mastectomy and axillary dissection will be randomized 1:1 into two groups: conventional fractionated (CF) radiotherapy of 50 Gy / 25 fractions and hypofractionated (HF) radiotherapy of 42.5 Gy/16 fractions, 5 fractions weekly.

The primary endpoint is loco-regional recurrence. Other cancer related events and acute/late radiation morbidities will also be evaluated. The patients will be followed for 10 years.

It is hypothesized that for women operated for high risk breast cancer with indication of postmastectomy adjuvant radiotherapy, hypofractionated radiotherapy is noninferior to conventional fractionated radiotherapy in terms of the efficacy and toxicities.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age18-75 years
* Pathologically confirmed invasive breast cancer
* Treated with mastectomy and axillary lymph node dissection with more than 10 resected lymph nodes. Immediate or delayed ipsilateral breast cancer reconstruction is accepted
* Negative surgical margins
* Pathologic T1-2N1 with at least one of the following risk factors: <40 years, Grade 3, lymphovascular invasion positive, ER/PR negative or HER2 overexpression, or pT3-4, or pN2-3 (four or more positive axillary lymph nodes)
* No distant metastases
* No supraclavicular or internal mammary nodes metastases
* ECOG:0-1
* Adjuvant systemic therapy with chemotherapy, endocrine therapy and anti-HER2 treatment is accepted.
* No neoadjuvant chemotherapy
* Fit for postoperative radiotherapy. No contraindications to radiotherapy
* Signed informed consent

Exclusion Criteria:

* Concurrent or previous malignancy excluding basal or squamous cell carcinoma of the skin
* Previous radiotherapy to the chest wall or regional lymph node areas
* Patients with severe non-malignant comorbidity in cardiovascular or respiration system
* Patients with medical contraindication for radiotherapy: systemic lupus erythematosus, cirrhosis
* pT1-2N1 with none of the following risk factors: <40 years, Grade 3, lymphovascular invasion positive, ER/PR negative or HER2 overexpression
* Patients with supraclavicular or internal mammary nodes metastases
* Known definitive clinical or radiologic evidence of metastatic disease
* Bilateral breast cancer or historically confirmed contralateral invasive breast cancer
* Treated with neoadjuvant chemotherapy
* ECOG: 3-4
* Pregnant or lactating
* Conditions indicating that the patient cannot go through the radiation therapy or follow up
* Unable or unwilling to sign informed consent

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1494 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
Loco-regional recurrence (LRR) | every 3 months during the first 2 years after the last fraction received, every 6 months during 3-5 years, every year during 6-10 years
  Defined as any clinical and biopsy-proven tumor recurrence involving the ipsilateral chest wall and/or regional nodes (including axillary, supraclavicular, infraclavicular, or internal mammary nodes). Time to loco-regional recurrence is defined as the interval starting from the date of randomization until the event. LRR will be assessed every 3 months during the first 2 years after the last fraction received, every 6 months during the following 3-5 years and every year thereafter through 10 years

SECONDARY OUTCOMES:
Distant metastasis free survival (DMFS) | every 3 months during the first 2 years after the last fraction received, every 6 months during 3-5 years, every year during 6-10 years
  Distant metastasis is defined as clinical detection of metastatic disease beyond the chest wall and/or regional lymph nodes or death or last visit. Distant metastasis free survival (DMFS) is defined as the interval starting from the date of randomization until to the event. Distant metastasis will be assessed every 3 months during the first 2 years after the last fraction received, every 6 months during the following 3-5 years and every year thereafter through 10 years.
Disease free survival (DFS) | every 3 months during the first 2 years after the last fraction received, every 6 months during 3-5 years, every year during 6-10 years
  Defined as the interval from the date of randomization to any disease recurrence or death or last visit. It will be assessed every 3 months during the first 2 years after the last fraction received, every 6 months during the following 3-5 years and every year thereafter through 10 years
Overall survival (OS) | every 3 months during the first 2 years after the last fraction received, every 6 months during 3-5 years, every year during 6-10 years
  Defined as the interval from the date of randomization to death or last visit. It will be assessed every 3 months during the first 2 years after the last fraction received, every 6 months during the following 3-5 years and every year thereafter through 10 years
CTCAE Toxicity Assessment-Acute toxicity | before treatment, every week of treatment, the end of treatment, 2 weeks, 3 months after the last fraction received, every year through 10 years
  Acute toxicity (development of radiation dermatitis, pruritus, pain, radiation esophagitis, and radiation pneumonitis) will be assessed according to toxicity criteria of CTCAE version 4.03 before treatment, every week of treatment, the end of treatment, 2 weeks, 3 months after the last fraction received and every year thereafter through 10 years
CTCAE Toxicity Assessment-Late toxicity | before treatment, every year after the last fraction received through 10 years
  Late toxicity (development of sclerosis in irradiated area and ischemic heart disease) will be assessed according to toxicity criteria of CTCAE version 4.03 before treatment and every year through 10 years following the completion of radiotherapy
LENT-SOMA Toxicity Assessment | before treatment, every year after the last fraction received through 10 years
  Development of dyspigmentation, telangiectasia in irradiated area and radiation pulmonary fibrosis will be assessed according to toxicity criteria of LENT-SOMA before treatment and every year through 10 years following the completion of radiotherapy
Number of patients with Arm Lymphedema | before treatment, every year after the last fraction received through 10 years
  Arm lymphedema defined as ≥10% increase in the treated arm circumference over baseline circumference compared to the contralateral arm. Arm circumference 15 cm above the medial epicondyle (upper arms) and 15 cm below the medial epicondyle (lower arms) will be measured before treatment and every year through 10 years following the completion of radiotherapy at every time point
Number of patients with impaired shoulder movement (Range of motion of the shoulders) | before treatment, every year after the last fraction received through 10 years
  Impaired shoulder movement is present when >20 degrees difference between arms at flexion and/or Abduction. Shoulder movement (Range of motion of the shoulders) will be assessed before treatment and every year through 10 years following the completion of radiotherapy
Number of patients with symptomatic rib fracture | before treatment, every year after the last fraction received through 10 years
  Symptomatic rib fracture will be diagnosed by evidence of a correlative lesion on plain film or CT. It will be assessed before treatment and every year through 10 years following the completion of radiotherapy
Number of patients with brachial plexopathy | before treatment, every year after the last fraction received through 10 years
  Brachial plexopathy will be documented if damage to the brachial plexus is suspected and patients have symptoms of pain, paresthesia, numbness, or other symptoms. Suspected cases of brachial plexopathy will be subject to confirmation by neurophysiological assessment. Brachial plexopathy will be assessed before treatment and every year through 10 years following the completion of radiotherapy
Number of patients with reconstruction complications | before treatment, every year after the last fraction received through 10 years
  For patients received mastectomy and reconstruction, the following complications will be assessed before treatment and every year through 10 years following the completion of radiotherapy: capsular contraction, partial or entire flap necrosis or loss, implant leakage and rupture, implant exposure, infection, hematoma/seroma and secondary surgical intervention
Cosmetic outcomes for patients received mastectomy with reconstruction | before treatment, every year after the last fraction received through 10 years
  The cosmetic outcomes will be evaluated by radiation oncologists, nurses and patients using digital photographs and Harvard/NSABP/RTOG Breast Cosmesis Grading Scale. Harvard/NSABP/RTOG Breast Cosmesis Grading Scale classifies the overall aesthetic results in four categories from excellent, good, fair to poor; comparing the reconstructed breast to the control breast. Excellent, there is minimal or no difference in the size or shape of the treated breast; good, slight difference in the size or shape of the treated breast; fair, obvious difference in the size or shape of the treated breast; and poor, marked change in the size or shape of the treated breast. The cosmetic outcomes will be assessed before treatment and every year through 10 years following the completion of radiotherapy. The breast cosmetic outcome will be measured by Harvard 4 scale (poor, fair, good, excellent) evaluation system
Quality of Life Life-EORTC QLQ-C30 (version 3) | before treatment, the end of treatment, every year after the last fraction received through 10 years
  Patients' quality of life will be assessed using self-administered questionnaire EORTC-QLQ-C30 (version 3) before treatment, the end of treatment, and every year through 10 years following the completion of radiotherapy
Quality of Life-EORTC breast-cancer module (BR23) | before treatment, the end of treatment, every year after the last fraction received through 10 years
  Patients' quality of life will be assessed using self-administered questionnaire EORTC breast-cancer module (BR23) before treatment, the end of treatment, and every year through 10 years following the completion of radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Jinli Ma, MD, PhD, Principal Investigator — Fudan University
Locations (3):
- China (3):
  - Suzhou Municipal hospital, Suzhou, Jiangsu
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Huangpu Branch, Shanghai ninth people's hospital, Shanghai, Shanghai Municipality